CLINICAL TRIAL: NCT01148940
Title: Sickle Cell Trait and the Risk of Venous Thromboembolism
Acronym: SCT&DVT
Status: Terminated | Type: Observational
Why Stopped: insufficent enrollment
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Henny Billett, Professor of Clinical Medicine and Pathology, Albert Einstein College of Medicine
Other Study IDs: 2009-539-001; 2009-539 (Other: IRB No.)
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Thrombosis
Keywords: sickle cell trait; thrombosis; D-Dimer
MeSH Terms: conditions — Thrombosis; Sickle Cell Trait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- White women with Hb AA: White pregnant and postpartum women with Hb AA
- Black women with Hb AA: Black pregnant and postpartum women with HbAA
- Black women with Sickle Trait: Black pregnant and postpartum women with HbAS

SUMMARY:
The purpose of this trial is to investigate D-Dimer levels, a surrogate marker of venous thromboembolism, in pregnant/postpartum white women as compared to pregnant/postpartum black women, and pregnant/postpartum women with sickle cell trait. The investigators will determine whether increased D-Dimer levels are reflected in a greater incidence of thrombosis in the postpartum patient, as well as the prevalence of symptomatic venous thrombosis in black patients as compared to pregnant white patients and women with sickle cell trait. The investigators will also investigate the effect of blood group on these parameters. If there is evidence that there is an increased risk of thrombosis in sickle cell trait, the investigators will plan a trial of prophylactic anticoagulation during the last trimester and the four weeks post partum for patients with sickle cell trait and compare this population to patients who do not receive prophylactic anticoagulation.

DETAILED DESCRIPTION:
Venous thromboembolism is the major cause of maternal mortality in the United States and there are emerging data that the thrombotic risk is higher in peripartum black women as compared to white women. The reasons are unclear: indeed, the few genetic risk factors for venous thrombosis that have been identified are more common in whites than blacks. This raises the possibility of yet undescribed mutations. To bolster this theory, some intriguing studies have noted a similar frequency of 'familial' thrombosis in blacks and whites, supporting the existence of yet unidentified hereditary component(s). Sickle cell anemia is a genetic disease more prevalent in the black population. Whereas sickle cell anemia has been associated with a prothrombotic state, there are limited data to support a prothrombotic state in sickle cell trait. We plan to examine whether sickle cell trait might play a role in increasing the incidence of thrombosis in the black population.

Peripartum women are 4-5 times more likely to develop venous thrombosis. Scant literature exists on the thrombotic risk in women from different races in the peripartum period and there are no studies evaluating venous thrombosis risk in sickle cell trait women during this time of increased thrombogenicity. In a retrospective analysis of deliveries of 12,000 women at Einstein/Montefiore, a higher incidence of venous thrombosis in black peripartum women was observed and, among the black population, a trend for sickle cell trait women to be at higher risk compared to black women with the normal hemoglobin (Hb) AA.

Given the medical importance and financial/sociological impact of venous thrombosis, it is important to determine whether black women, and specifically black women with sickle cell trait, are really at increased risk for thromboembolic disease during the peripartum period and, if so, what intervention(s) might mitigate this risk. We propose to perform a prospective study investigating peripartum white Hb AA, black Hb AA, and black sickle cell trait women by assessing D-Dimer levels. The D-Dimer levels will be assayed at defined times during the peripartum and correlated with pregnancy complications, as well as neonatal and birth data, thrombosis and, in selected cases, lower extremity duplex ultrasonography. If, after analysis, there is evidence confirming an increased thrombotic risk, we will design and institute an interventional trial. The purpose of this application is to fill in the gaps of current knowledge regarding the role of race in venous thromboembolism, to test different methodologies for studying this significant health problem, and to lay the groundwork for clinical trial development to determine whether therapeutic intervention with prophylactic anticoagulation is beneficial during the peripartum period for patients with sickle cell trait.

ELIGIBILITY:
Inclusion Criteria:

* Peripartum women (White, Black) with Hemoglobin AA or AS

Exclusion Criteria:

* Hispanic ethnicity

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women who are pregnant or postpartum
Study Population: Pregnant and postpartum women
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henny H Billett, MD MSc, Principal Investigator — Albert Einstein College of Medicine/Montefiore Medical Ctr
Locations (1):
- Montefiore Medical Center (Einstein), The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plans at present

RESULTS

PARTICIPANT FLOW:
Groups:
- White Women With HbAA: White pregnant and post partum women with Hb AA
- Black Women With Hb AA: Black pregnant and post partum women with HbAA
- Black Women With SCT: Black pregnant and postpartum women with HbAS
Period: Overall Study
Arm/Group | White Women With HbAA | Black Women With Hb AA | Black Women With SCT
Started | 7 | 27 | 0
Completed | 7 | 27 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- White; Black: self-described
- Total: Total of all reporting groups
Arm/Group | White | Black | Total
Number analyzed (Participants) | 7 | 27 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 27 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29.3 [18.2 to 39.1] | 29.3 [18.2 to 39.1] | 29.3 [18.2 to 39.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 27 | 34
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 27 | 34

OUTCOME MEASURES:

1. Primary Outcome: D-Dimer Levels Than in Black Women With Hb AA and White Women With Hb AA.
Description: High D-Dimer levels are regarded as potentially prothrombotic markers and are often elevated in pregnancy and the postpartum. There are some data to suggest that sickle cell trait may also be prothrombotic.To investigate whether D-Dimer levels are higher in black peripartum women with SCT than in black or white pregnant/postpartum patients who have Hb AA, we will measure the D-Dimer, on a continuous scale, in the pregnant/postpartum population of each group. It is known that D-Dimer levels >1.0 mg/ml may be predictive of increased thrombotic risk. We will compare mean D-Dimer of Black SCT women, Black AA women and White AA women to determine whether higher D-Dimer levels, which may be a measure of hypercoagulability, are higher in women with SCT.
Time Frame: Date of delivery until 4-5 weeks postpartum.
Population: did not recruit any women with sickle cell trait
Measure: Mean (95% Confidence Interval); unit: micrograms/ml
Groups:
- White Women With HbAA: White women pregnant and postpartum with HbAA
- Black Women With HbAA: Black women pregnant and postpartum with HbAA
- Black Women With SCT: Black women pregnant and postpartum with HbAS
Arm/Group | White Women With HbAA | Black Women With HbAA | Black Women With SCT
Number analyzed (Participants) | 7 | 27 | 0
micrograms/ml | 1.370 [.773 to 1.853] | 1.850 [1.515 to 4.185] |

ADVERSE EVENTS:
Time Frame: Blood was collected on day 7-10 post delivery and again at 4 weeks post partum. Total duration was therefore about 4-5 weeks. Study duration was July 2010 - June 2011
Description: The only potential adverse events were the 1) potential for the inadvertent release of protected health information and 2) the risks of venipuncture including local ecchymoses and rarely, syncope. Neither of these adverse events occurred. The only group were there were 0 potentially at risk was the SCT group - that is because no SCT patients were in the study.
Groups:
- White Women With HbAA: White pregnant/postpartum women with HbAA
- Black Women With HbAA: black pregnant/postpartum women with HbAA
- Black Women With SCT: black women with HbAS
Arm/Group | White Women With HbAA | Black Women With HbAA | Black Women With SCT
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/27 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/27 | 0/0
Other Adverse Events (participants affected / at risk) | 0/7 | 0/27 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No